CLINICAL TRIAL: NCT04028336
Title: The Strategy of "Pulmonary Opening by Titration of Positive End-expiratory Pressure" Means of a Pulmonary Recruitment Maneuver in Patients With Acute Respiratory Distress Syndrome: for Which Patients?
Acronym: OPPRED
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Technical difficulties
Sponsor: Centre Hospitalier de Lens (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: PI2019-01/OPPRED/DRMARC
Record Dates: First submitted 2019-07-09; First posted 2019-07-22 (Actual); Last update posted 2021-03-04 (Actual); Status verified 2021-03

CONDITIONS: Respiratory Distress Syndrome, Adult
MeSH Terms: conditions — Respiratory Distress Syndrome

STUDY DESIGN:
Intervention Model Description: All patients in intensive care and severe, moderate ARDS will be included in this study. All patients will benefit from Lung ultrasound (LUS) with a mapping of each lung looking for normal or pathological lung profiles, as well as a measurement of esophageal pressure (Peso) at rest. A "PEP titration pulmonary opening" (PEP-OP) test using a recruitment maneuver was then performed in all patients followed by a new LUS and Peso measurement.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- TITRATION (Experimental): All patients hospitalized in intensive care and meeting inclusion criteria and without criteria for non-inclusion will be included in this study. All patients will benefit from Lung ultrasound (LUS) and esophageal pressure measurement (Peso) according to the habits of the service. A "PEP titration pulmonary opening" (PEP-OP) test using a recruitment maneuver was then performed in all patients followed by a new LUS and Peso measurement.
  Interventions: Other: TITRATION

INTERVENTIONS:
Other: TITRATION — PEP titration pulmonary opening (PEP-OP) was performed in all patients followed by new LUS and Peso measurement.

SUMMARY:
Pulmonary recruitment maneuvers open these lung areas and appropriate adjustment of positive expiratory pressure (PEP) helps to stabilize recruitment and reduce the stress associated with alveolar opening and closing. Its beneficial effects in the lung affected by Acute Respiratory Distress Syndrome (ARDS) remain unclear. The hypothesis is that there is a heterogeneous effect of the recruitment maneuver according to the phenotype of ARDS. It is important to be able to define responder patients from non-responders to this recruiting maneuver.

DETAILED DESCRIPTION:
It will be a prospective interventional study in resuscitation patients with severe or moderate ARDS. This study will be multicentric between the University Hospital of Amiens and intensive care of Lens, intensive care of Bethune and intensive care of Arras. All patients in intensive care and severe, moderate ARDS will be included in this study. All patients will benefit from Lung ultrasound (LUS) with a mapping of each lung looking for normal or pathological lung profiles, as well as a measurement of esophageal pressure (Peso) at rest. A "PEP titration pulmonary opening" (PEP-OP) test using a recruitment maneuver was then performed in all patients followed by a new LUS and Peso measurement.

ELIGIBILITY:
Inclusion Criteria:

Will be included in the study, patients:

* Major patient (age ≥18 years)
* Controlled assisted ventilation, sedation and curarization adapted to the respirator.
* Within the first 72 hours of an ARDS (PaO2 / FiO2 ≤ 200 mmHg, FiO2 ≥ 60% and PEEP of ≥5 cmH20) (as recommended by the Berlin criteria)
* Decision of intensivist in charge of the patient to put an oesophageal probe
* After hemodynamic optimization (evaluation of the preload dependence and need for catecholamines)
* Decision of the intensivist in charge of the patient to perform a pulmonary opening test by titration of PEEP by means of a pulmonary recruitment test.

Exclusion Criteria:

* Patients under the age of 18
* Pregnant women, women who are parturient or breastfeeding
* Patients with pulmonary broncho-emphysematous pathology or at risk of presenting it.
* Patients with a history of barotrauma or at risk of presenting it.
* Patients with a history of intracranial hypertension
* Patients with suspected or proven right ventricular dysfunction or uncontrolled hemodynamic instability after hemodynamic management.
* Patients with a contraindication to the placement of an oesophageal tube (esophageal surgery, severe esophageal pathology)
* Patients under guardianship or curatorship or deprived of liberty.
* Patients who are legally protected
* Patient not covered by French national health insurance

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 4 (Actual)
Dates: Start 2019-12-20 (Actual); Primary Completion 2021-01-07 (Actual); Study Completion 2021-01-07 (Actual)

PRIMARY OUTCOMES:
oxygenation and pulmonary compliance | at 1 hours of the PEP-OP test.
  The primary outcome is oxygenation (PaO2 / FiO2) and pulmonary compliance ((Pplat-Pep) / VT) at 1h of the PEP-OP test.

SECONDARY OUTCOMES:
Oxygenation (PaO2 / FiO2) at 6h, 12h, 24h | at 6 hours, 12 hours, 24 hours of the PEP-OP test
  Oxygenation (PaO2 / FiO2) at 6h, 12h, 24h
Mechanical ventilation time | Discharge from intensive care unit
  Mechanical ventilation time
Hospitalization in intensive care time | Discharge from intensive care unit
  Hospitalization in intensive care time
The need for recourse to alternative therapies of oxygenation | Discharge from intensive care unit
  The need for recourse to alternative therapies of oxygenation
Incidence of barotrauma | After PEP-OP
  Incidence of barotrauma
Pulmonary compliance at 6 hours, 12 hours and 24 hours | at 6 hours, 12 hours and 24 hours of the PEP-OP test.
  Pulmonary compliance at 6 hours, 12 hours and 24 hours

CONTACTS AND LOCATIONS:
Overall Officials: Julien MARC, DR, Principal Investigator — Hospital of Lens
Locations (4):
- France (4):
  - Chu Amiens, Amiens
  - CH Arras, Arras
  - Ch Germon Et Gauthier, Béthune
  - Hospital Dr Schaffner, Lens